CLINICAL TRIAL: NCT00907413
Title: Photodynamic Therapy for Palliation of Unresectable Cholangiocarcinoma A Multicenter, Open Label, Randomized, Controlled Phase III Trial
Brief Title: Photodynamic Therapy (PDT) Trial for Palliation of Cholangiocarcinoma
Acronym: PDT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI relocated and reopened trial in new university
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief of Endoscopy, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13898
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Cholangiocarcinoma
Keywords: cancer; bile duct
MeSH Terms: conditions — Cholangiocarcinoma; Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERCP and PDT (Experimental): Endoscopic Retrograde Cholangio Pancreatography (ERCP) and stenting combined with Photodynamic Dynamic Therapy ERCP and PDT
  Interventions: Procedure: ERCP and Photodynamic Therapy; Procedure: ERCP only
- ERCP alone (Active Comparator): Endoscopic Retrograde Cholangio Pancreatography (ERCP) with stenting alone
  Interventions: Procedure: ERCP only

INTERVENTIONS:
Procedure: ERCP and Photodynamic Therapy — Photodynamic Therapy is a new therapeutic approach that specifically targets neoplastic cells. This therapy has been used in other tumors as a local treatment and involves the intravenous administration of a photosensitizing agent followed by activation of the agent by illumination with non-thermal light of a specific wavelength, resulting in cell death from direct cytotoxicity and ischemic necrosis. Cytotoxicity is directly proportional to tissue oxygenation.
  Arms: ERCP and PDT
Procedure: ERCP only — Endoscopic retrograde cholangiopancreatography and stenting.

SUMMARY:
This research study is a phase III double arm, multicenter, randomized controlled clinical trial comparing endoscopic retrograde cholangiopancreatography (ERCP) and stenting plus photodynamic therapy (PDT) versus ERCP with stenting alone in adult patients with unresectable cholangiocarcinoma.

The study objectives are to investigate the efficacy of photodynamic therapy (PDT) in increasing the survival time of patients with unresectable cholangiocarcinoma and to assess the effect of PDT on both cholestasis and health-related quality of life (HRQoL).

DETAILED DESCRIPTION:
The study objectives are to investigate the efficacy of photodynamic therapy (PDT) in increasing the survival time of patients with unresectable cholangiocarcinoma and to assess the effect of PDT on both cholestasis and health-related quality of life (HRQoL).

ELIGIBILITY:
Inclusion Criteria:

* Patient is age 18 years or older
* Patient is diagnosed with non-resectable cholangiocarcinoma, as determined by CT within 30 days of enrollment and CT shows Bismuth Tumor Stage as: IIIa, IIIb, IV (Bismuth tumor stage I and II are not eligible to participate)
* Patients must have adequate organ and marrow function as defined below:

  * Patient's INR ≤ 2 within 30 days of treatment
  * Patient's platelets > 50,000/cmm within 30 days of treatment
  * Patient's Absolute Neutrophil Count (ANC) > 1,500/cmm within 30 days of treatment
  * Patient's creatinine ≤ 3 mg/dL within 30 days of treatment
* Patient has the ability to understand and the willingness to comply with the study procedures and provide written informed consent to participate in the study

Exclusion Criteria:

* Patient was diagnosed with cholangiocarcinoma more than 3 months ago
* Patient has any metastatic disease
* Patient has acute porphyria
* Subjects exhibiting neurologic or cutaneous symptoms will undergo urinary delta-aminolevulinic acid and porphobilinogen dosage tests to determine severity.
* Patient is pregnant (Women of child bearing age must have a negative pregnancy test prior to registration and must agree to use adequate contraception during study therapy)
* Patient has a concurrent non solid malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Survival time in each group will be compared as well as effect of each treatment arm on cholestasis and HRQoL | 2.4 years

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlotteville, Virginia, United States

REFERENCES:
- [Derived] Cerecedo-Rodriguez J, Phillips M, Figueroa-Barojas P, Kumer SC, Gaidhane M, Schmitt T, Kahaleh M. Self expandable metal stents for anastomotic stricture following liver transplant. Dig Dis Sci. 2013 Sep;58(9):2661-6. doi: 10.1007/s10620-013-2703-0. Epub 2013 May 24. PMID 23703448